CLINICAL TRIAL: NCT06167941
Title: Identification of Integrin ab Expression in Lung Cancer Patients for Clinical Application of Cancer-Target Fluorescent Contrast Agent for Image-Induced Precise Lung Cancer Surgery
Brief Title: Identification of Integrin ab Expression in Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, MD, Korea University Guro Hospital
Other Study IDs: 2019GR0460
Record Dates: First submitted 2023-11-20; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Expression of Integrin ανβ3 in Lung Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — tissue slide of lung cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung cancer: adenocarcinoma and squamous carcinoma
  Interventions: Biological: Lung cancer types

INTERVENTIONS:
Biological: Lung cancer types — Cancer tissue matched to normal tissue, all from the same patient

SUMMARY:
It has been reported that the expression rates of integrin αvβ3 and integrin αvβ5 in NSCLC are 89% and 100%, respectively. Among RGD (Arg-Gly-Asp) peptides, cRGDyK peptide (cRGD) known as integrin ανβ3 and ανβ5 antagonist has been widely used for targeting various cancers including NSCLC, glioblastoma, and colon carcinoma as well as prostate cancer. In this study, the investigators aim to analysis the expression of integrin ανβ3 in lung cancer patients.

DETAILED DESCRIPTION:
Patient samples: From the Human Resource Bank of the Institute of Pathology, Korea University, the investigators collected paraffin-embedded tissue sections from 61 patients with NSCLC (adenocarcinoma =50, squamous cell carcinoma = 11) who had undergone surgical treatment for NSCLC at Korea University Guro Hospital between 2015 and 2018 under the IRB of Guro Hospital 2019GR0460. Samples were excluded when patients had undergone perioperative chemo- or radiotherapy. Among the tissues excised from lung cancer patients, lung cancer and normal tissue were classified as pathologically, defined as normal tissue and cancer tissue, and stained with an integrin ανβ3 primary antibody.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC (adenocarcinoma or squamous cell carcinoma) who had undergone surgical treatment for NSCLC at Korea University Guro Hospital between 2015 and 2018

Exclusion Criteria:

* patients had undergone perioperative chemo- or radiotherapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC (adenocarcinoma or squamous cell carcinoma) who had undergone surgical treatment for NSCLC at Korea University Guro Hospital between 2015 and 2018
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
integrin expression level | 20 months
  Integrins expression level categorized to high and low

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Koo Kim, Study Director — Korea University Guro Hospital
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided